CLINICAL TRIAL: NCT01945580
Title: A Prospective, Non-Randomized, Parallel Cohort, Multi-Center Study of Xenform vs. Native Tissue for the Treatment of Women With Anterior/Apical Pelvic Organ Prolapse
Brief Title: Xenform Postmarket Surveillance Study
Acronym: Xenform
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U9920; AUGS PFD Outcome Registry (Registry Identifier: AUGS PFD Outcome Registry)
Record Dates: First submitted 2013-09-15; First posted 2013-09-18 (Estimated); Results first posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-03

CONDITIONS: Pelvic Organ Prolapse
Keywords: POP; Transvaginal; Native Tissue Repair; Repair Augmented with Mesh; Biologic Graft; Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Xenform (Active Comparator): Prolapse Repair with Xenform Soft Tissue Repair Matrix
  Interventions: Procedure: Prolapse Repair
- Control (Active Comparator): Prolapse Repair with Native Tissue Only
  Interventions: Procedure: Prolapse Repair

INTERVENTIONS:
Procedure: Prolapse Repair — Transvaginal anterior/apical pelvic organ prolapse repair
  Other Names: Transvaginal; Prolapse; POP Repair; Anterior; Apical

SUMMARY:
To compare transvaginal repair with a biologic graft to traditional native tissue repair in women surgically treated for anterior and/or apical pelvic organ prolapse.

DETAILED DESCRIPTION:
The primary objective is to evaluate clinical effectiveness of transvaginal repair with Xenform against traditional native tissue repair in women surgically treated for anterior and/or apical pelvic organ prolapse. Secondary objectives are to evaluate Xenform-related complications and subject reported outcomes.

The primary endpoint of the study is to achieve non-inferiority of transvaginal repair with Xenform over native tissue repair at 36 months as compared to baseline. Success will be based on a composite of objective and subjective measures.

Additionally, a co-primary endpoint of the study is to achieve non-inferiority of transvaginal repair with Xenform to native tissue repair for safety by comparing rates of serious device or serious procedure related complications between baseline and the 36 month time point.

The secondary endpoints of the study include assessments of complications and subject reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Subject is female
* Subject is at least 18 years of age
* Subject has pelvic organ prolapse with the leading edge at or beyond the hymen. At or beyond the hymen is defined as POP-Q scores of Ba≥0 (for prolapse of the anterior compartment alone) or C≥0 (for prolapse of the apical compartment alone) or C≥-1/2 TVL and Ba≥0 (for a multi-compartment prolapse that includes the anterior and apical compartments).
* Subject reports a bothersome bulge they can see or feel per PFDI-20, question 3, response of 2 or higher (i.e., responses of "somewhat", "moderately", or "quite a bit")
* Subject or subject's legally authorized representative is willing to provide written informed consent
* Subject is willing and able to comply with the follow-up regimen

Exclusion Criteria:

* Subject is pregnant or intends to become pregnant during the study
* Subject has an active or chronic systemic infection including any gynecologic infection, untreated urinary tract infection (UTI) or tissue necrosis
* Subject has history of pelvic organ cancer (e.g. uterine, ovarian, bladder, colo-rectal or cervical)
* Subject has had prior or is currently undergoing radiation, laser therapy, or chemotherapy in the pelvic area
* Subject has taken systemic steroids (within the last month), or immunosuppressive or immunomodulatory treatment (within the last 3 months)
* Subject has systemic connective tissue disease (e.g. scleroderma, systemic lupus erythematosus (SLE), Marfan syndrome, Ehlers Danlos, collagenosis, polymyositis, polymyalgia rheumatica)
* Subject has chronic systemic pain that includes the pelvic area or chronic focal pain that involves the pelvis
* Subject has uncontrolled diabetes mellitus (DM)
* Subject has a known neurologic or medical condition affecting bladder function (e.g., multiple sclerosis, spinal cord injury or stroke with residual neurologic deficit)
* Subject is seeking obliterative vaginal surgery as treatment for pelvic organ prolapse (colpocleisis)
* Subject is not able to conform to the modified dorsal lithotomy position
* Subject is currently participating in or plans to participate in another device or drug study during this study
* Subject has a known sensitivity to any Xenform component
* Subject has had previous prolapse repair with mesh in the target compartment
* Subject is planning to undergo a concomitant prolapse repair with use of mesh in the non-target compartment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2014-02-10 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rosenblatt, MD, Principal Investigator — Mount Auburn Hospital
Locations (25):
- United States (25):
  - University of California, Irvine Medical Center, Orange, California
  - Emory Hospital, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Cherokee Womens Health Specialist, Canton, Georgia
  - NorthShore University Health System, Skokie, Illinois
  - Acadia Women's Health, Crowley, Louisiana
  - Chesapeake Urology Research Associates, Hanover, Maryland
  - Chesapeake Urology Research Associates, Owings Mills, Maryland
  - Mount Auburn Hospital, Cambridge, Massachusetts
  - Beyer Research, Kalamazoo, Michigan
  - Cooper University Hospital, Voorhees Township, New Jersey
  - University of Buffalo, Buffalo, New York
  - Beth Israel Medical Center, New York, New York
  - NYU Langone Medical Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Carolina Urology Partners, Gastonia, North Carolina
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - Prime Care of SEO, Dresden, Ohio
  - Prisma Health System, Greenville, South Carolina
  - Southern Urogynecology, West Columbia, South Carolina
  - Center for Pelvic Health, Franklin, Tennessee
  - Practice Research Organization, Dallas, Texas
  - Houston Metro Urology, Houston, Texas
  - Las Colinas ObGyn, Irving, Texas
  - MultiCare Women's Health Care, Covington, Washington

REFERENCES:
- [Derived] Lipetskaia L, Gonzalez RR, Wu JM, Northington GM, Henley BR, Lane F, Brucker BM, Jarnagin B, Rosenblatt PL. Thirty-six-month Prospective Study of Transvaginal Bovine Graft vs Native Tissue Repair for the Treatment of Pelvic Organ Prolapse. Urology. 2022 Sep;167:234-240. doi: 10.1016/j.urology.2022.06.003. Epub 2022 Jun 15. PMID 35716871

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 412 subjects were screened and 374 subjects were enrolled in the Xenform Postmarket Surveillance Study. 228 subjects were enrolled into the Xenform arm and 146 subjects into the NTR arm. 339 subjects from the AUGS PFD Registry (64 subjects from BSC's Uphold™ LITE 522 study [NCT01917968], 69 subjects from Acell's MatriStem® 522 study & 206 subjects from Coloplast's 522 Restorelle® study) were pulled into the NTR arm for a total of 485 subjects in the NTR cohort and a total of 713 subjects overall
Period: Overall Study
Arm/Group | Xenform | Control
Started | 228 | 485
Completed | 176 | 401
Not Completed | 52 | 84
Not completed — Withdrawal by Subject | 13 | 35
Not completed — Physician Decision | 3 | 2
Not completed — Lost to Follow-up | 26 | 39
Not completed — Death | 7 | 2
Not completed — Patient moved out of state | 0 | 1
Not completed — Moved out of state and firmly desired to withdraw. AE still not recovered and not resolved. | 1 | 0
Not completed — Family illness - unable to return | 0 | 1
Not completed — Weather emergency at time visit due; per sponsor completed study due to being too far out of window | 0 | 1
Not completed — Death in family, then rescheduled but considered too far out of window to bring back | 0 | 1
Not completed — Noncompliance with 36 month visit | 1 | 0
Not completed — The patient moved. | 1 | 0
Not completed — No data available | 0 | 2

BASELINE CHARACTERISTICS:
Population: 412 subjects were screened and 374 subjects were enrolled in the Xenform Postmarket Surveillance Study. 228 subjects were enrolled into the Xenform arm and 146 subjects into the NTR arm. 339 subjects from the AUGS PFD Registry (64 subjects from BSC's Uphold™ LITE 522 study, 69 subjects from Acell's MatriStem® 522 study and 206 subjects from Coloplast's 522 Restorelle® study) were pulled into the NTR arm for a total of 485 subjects in the NTR cohort and a total of 713 study subjects overall.
Groups:
- Total: Total of all reporting groups
Arm/Group | Xenform | Control | Total
Number analyzed (Participants) | 228 | 485 | 713
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (12.7) | 61.8 (10.5) | 60.7 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 228 | 485 | 713
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 20 | 47
  Not Hispanic or Latino | 199 | 457 | 656
  Unknown or Not Reported | 2 | 8 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 11 | 17
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 16 | 55 | 71
  White | 198 | 409 | 607
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 9 | 16
Region of Enrollment [Number; unit: participants]
  United States | 228 | 485 | 713
Smoking [Count of Participants; unit: Participants]
  Current | 21 | 38 | 59
  Previous | 41 | 139 | 180
  Never | 164 | 308 | 472
  Not Recorded | 2 | 0 | 2
Diabetes [Count of Participants; unit: Participants] | 22 | 63 | 85
Menopausal Status [Count of Participants; unit: Participants]
  Premenopausal | 39 | 54 | 93
  Perimenopausal | 19 | 27 | 46
  Postmenopausal | 170 | 404 | 574
Previous Pelvic Surgery [Count of Participants; unit: Participants] | 136 | 235 | 371

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Success at 36 Months
Description: The primary endpoint of the study was to achieve non-inferiority of transvaginal repair with Xenform over NTR at 36 months as compared to baseline. Success was based on a composite of objective and subjective measures.
  1. Subjective success was achieved if the patient denied symptoms of vaginal bulging per Pelvic Floor Distress Inventory (PFDI-20) question 3, answering "no" or "yes" but "Not at all" bothersome (< 2).
  2. Anatomic success (in the operated compartment):
     * Anterior segment: Leading edge of anterior prolapse was at or above the hymen or Pelvic Organ Prolapse Quantification System (POP-Q) point Ba ≤ 0.
     * Apical segment: The vaginal apex did not descend more than one-half into the vaginal canal (i.e., POP-Q point C < -1/2 TVL) for multi-compartment prolapse or POP-Q point C ≤ 0 for single compartment apical prolapse.
  3. No retreatment for POP: no additional surgical treatment for POP in the segment(s) of the vagina treated at the index surgery or no pessary use
Time Frame: 36 Months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Xenform | Control
Number analyzed (Participants) | 228 | 485
Participants | 191 | 390
Statistical Analysis 1: Comparison: Xenform vs Control; Test type: Non-Inferiority — With type I error of 0.05 and type II error of 0.20 (power 80%), 362 subjects (181 subjects per arm) are needed to detect non-inferiority of transvaginal biologic to native tissue repair, using a margin of 12.0%; Adjusted Difference in Percentages = 0.2, 90% CI 2-sided [-5.6 to 5.9] — The propensity adjusted treatment difference of Xenform transvaginal mesh (TVM) minus NTR was estimated and missing data was handled using multiple imputation method

2. Primary Outcome: Number of Participants With One or More Serious Device-related and/or Procedure-Related Adverse Events
Description: Co-primary endpoint of the study was to achieve non-inferiority of transvaginal mesh repair with Xenform to NTR for safety by comparing rates of serious device-related or serious procedure-related complications between baseline and the 36-month time point.
Time Frame: 36 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Xenform | Control
Number analyzed (Participants) | 228 | 485
Participants | 12 | 13
Statistical Analysis 1: Comparison: Xenform vs Control; Test type: Non-Inferiority — With type I error of 0.05 and type II error of 0.10 (power 90%), 308 subjects (154 subjects per arm) are needed to detect non-inferiority with a margin of 11.6%; Adjusted Difference in Percentages = 2.0, 90% CI 2-sided [-0.8 to 4.7] — The propensity score adjusted difference in SAE rate of Xenform transvaginal mesh (TVM) vs. NTR was estimated

3. Secondary Outcome: Number of Participants With Mesh Erosion
Description: Incidence of Mesh Erosion at 36 months
Time Frame: 36 months
Population: The population includes the 228 subjects in the Xenform arm of the study.
Measure: Count of Participants; unit: Participants
Groups:
- Total: Inclusive
- Mild; Moderate; Severe: Measure of Severity
Arm/Group | Total | Mild | Moderate | Severe
Number analyzed (Participants) | 228 | 228 | 228 | 228
Participants | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Mesh Exposure
Description: Incidence of mesh exposure at 36 months
Time Frame: 36 Months
Population: The population includes the 228 subjects in the Xenform arm of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Total | Mild | Moderate | Severe
Number analyzed (Participants) | 228 | 228 | 228 | 228
Participants | 2 | 2 | 0 | 0

5. Secondary Outcome: Number of Participants With de Novo Dyspareunia
Description: Incidence of de novo dyspareunia at 36 months
Time Frame: 36 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Xenform | Control
Number analyzed (Participants) | 228 | 485
Participants | 2 | 6

6. Secondary Outcome: Subject Specific Outcomes Measured With the Pelvic Floor Impact Questionnaire (PFIQ-7)]
Description: Improvement in subject specific outcomes at 36 months compared to baseline [quality of life (QOL) per the Pelvic Floor Impact Questionnaire (PFIQ-7)]
  The PFIQ-7 is composed of three separate but related assessments: the UIQ-7 addresses the impact of urinary incontinence symptoms, the CRAIQ-7 addresses the impact of colorectal-anal or bowel symptoms, and the POPIQ-7 addresses impact of vaginal and pelvic symptoms. For each question, the low score (0) corresponds to "not at all" and the high score (3) corresponds to "quite a bit". The scores for the UIQ-7, CRAIQ-7 and POPIQ-7 are additive to yield the final PFIQ-7 score. The scale scores are then added together to get the total PFIQ-7 score, which ranges from 0-300. A lower score means there is a lesser effect on quality of life.
  Reported score is change from baseline at 36 months.
Time Frame: 36 months
Population: The 174 Xenform arm participants and 399 Native Tissue Repair arm participants are indicative of the available information at the 36 month timepoint (i.e. the number of participants who completed the PFIQ-7 questionnaire at Baseline and 36 months).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Xenform | Control
Number analyzed (Participants) | 174 | 399
score on a scale | -55.2 (62.8) | -41.9 (55.0)

7. Secondary Outcome: Subject Specific Outcomes Measured by the Pelvic Floor Symptoms Per the Pelvic Floor Distress Inventory (PFDI-20)
Description: Improvement in subject specific outcomes at 36 months compared to baseline [pelvic floor symptoms per the Pelvic Floor Distress Inventory (PFDI-20)]
  The Pelvic Floor Distress Inventory-20 (PFDI-20) is complimentary to the PFIQ-7 and focuses on symptoms of distress in the same compartmentalized fashion as the PFIQ-7. Like the PFIQ-7, the PFDI-20 consists of three components: Urinary Distress Inventory (UDI; 6 questions), the Pelvic Organ Prolapse Distress Inventory (POPDI; 6 questions), and Colorectal-Anal Distress Inventory (CRADI; 8 questions). The scoring for the PFDI-20 is similar to the PFIQ-7 where each individual component score is summed. The total ranges from 0 to 300 with a higher score indicating a greater impact to QOL (i.e., distress symptoms are more noticeable) and a lower score indicating a lesser impact to QOL (i.e., distress symptoms are less noticeable).
  The reported result is change from baseline at 36 months.
Time Frame: 36 months
Population: The 175 Xenform arm participants and 400 Native Tissue Repair arm participants are indicative of the available information at the 36 month timepoint (i.e. the number of participants who completed the PFDI-20 questionnaire at Baseline and 36 months).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Xenform | Control
Number analyzed (Participants) | 175 | 400
score on a scale | -80.8 (58.6) | -77.2 (56.1)

8. Secondary Outcome: Subject Specific Outcomes Measured by the Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ-12)
Description: Improvement in subject specific outcomes at 36 months compared to baseline [change in sexual functioning per the Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ-12)]
  This is a self-administered questionnaire and the responses are graded on a five-point Likert scale ranging from 0 (always) to 4 (never). Values range from 0 to 48 and a higher score indicates better sexual function.
  The reported result is change from baseline at 36 months.
Time Frame: 36 months
Population: The 78 Xenform arm participants and 156 Native Tissue Repair arm participants are indicative of the available information at the 36 month timepoint (i.e. the number of participants who completed the PISQ-12 questionnaire at Baseline and 36 months).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Xenform | Control
Number analyzed (Participants) | 78 | 156
score on a scale | 5.0 (7.2) | 4.3 (5.8)

9. Secondary Outcome: Subject Specific Outcomes: Pain Measured by the TOMUS Pain Scale
Description: Improvement in subject specific outcomes at 36 months compared to baseline [pain per the TOMUS pain scale]
  The TOMUS Pain Score, a visual analog instrument with a scale of 0 (no pain sensation) to 10 (most intense pain sensation imaginable), was used to assess pain associated with surgery for pelvic organ prolapse in this study. There are seven (7) questions each with a maximum score of 10 and a possible score range of 0-70).
  The reported results are change from baseline at 36 months.
Time Frame: 36 months
Population: The 175 Xenform arm participants and 399 Native Tissue Repair arm participants are indicative of the available information at the 36 month timepoint (i.e. the number of participants who completed the TOMUS pain scale at Baseline and 36 months).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Xenform | Control
Number analyzed (Participants) | 175 | 399
score on a scale | -4.8 (8.8) | -4.0 (8.3)

10. Secondary Outcome: Subject Improvement Measured by the Patient Global Impression of Improvement for Prolapse (PGI-I)
Description: Assessment of subject's level of improvement, measured by the Patient Global Impression of Improvement for Prolapse (PGI-I)
  The Patient Global Impression of Improvement (PGI-I) for prolapse symptoms is a validated QOL instrument that assesses patient perception of overall improvement after surgical interventions for POP.12 The scale rates the patient's improvement or worsening of prolapse symptoms relative to baseline. The scale is as follows: 1- Very much better; 2- Much better; 3- A little better; 4- No change; 5- A little worse; 6- Much worse; 7- Very much worse. Assessments were performed at 6-month intervals beginning 6 months after the index procedure.
Time Frame: 36 months
Population: The 175 Xenform arm participants and 399 Native Tissue Repair arm participants are indicative of the available information at the 36 month timepoint (i.e. the number of participants who completed the PGI-I at Baseline and 36 months).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Xenform | Control
Number analyzed (Participants) | 175 | 399
score on a scale | 1.6 (0.9) | 1.4 (0.9)

11. Secondary Outcome: Number of Participants With Re-Intervention or Re-Surgery
Description: Absence of re-intervention or re-surgery for recurrence or persistence of POP or Xenform exposure/erosion
Time Frame: 36 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Xenform | Control
Number analyzed (Participants) | 228 | 485
Participants
  Office-Based Intervention for Recurrent Prolapse | 1 | 2
  Surgical Intervention for Recurrent Prolapse | 5 | 15
  Office-Based Intervention for Complications | 23 | 40
  Surgical Intervention for Complications | 15 | 34

12. Secondary Outcome: Surgical Success
Description: Surgical success based on the following composite outcome:
  1. Subjective success: Patient denied symptoms of vaginal bulging per PFDI-20 question 3, answering "no" or "yes" but "Not at all" bothersome (˂ 2)
  2. Anatomic success (in the operated compartment):
     * Anterior Segment: No anterior prolapse at or beyond the hymen or POP-Q point Ba ˂ 0
     * Apical Segment: The vaginal apex did not descend more than one-half into the vaginal canal (i.e., POP-Q point C ˂ 1/2 TVL) for multi-compartment prolapse or POP-Q point C ˂ 0 for prolapse of the apical compartment alone
     * No retreatment for POP (treated segment): No additional surgical treatment for POP in the segment(s) of the vagina treated at the index surgery or no pessary use since index surgery ('treated segment' refers to the target compartments in this study, which are the anterior and apical compartments)
Time Frame: 36 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Xenform | Control
Number analyzed (Participants) | 228 | 485
Participants | 183 | 351

13. Secondary Outcome: Incidence of Complications
Description: Incidence of the following device-related or procedure-related adverse events (AEs): pelvic pain, infection, vaginal shortening, atypical vaginal discharge, neuromuscular problems, vaginal scarring, de novo vaginal bleeding, fistula formation and/or de novo voiding dysfunction.
Time Frame: 36 Months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Xenform | Control
Number analyzed (Participants) | 228 | 485
Participants
  pelvic pain | 14 | 28
  infection | 25 | 68
  vaginal shortening | 0 | 0
  atypical vaginal discharge | 2 | 3
  neuromuscular problems | 3 | 14
  vaginal scarring | 3 | 1
  de novo vaginal bleeding | 3 | 7
  fistula formation | 0 | 0
  de novo voiding dysfunction | 35 | 23

ADVERSE EVENTS:
Time Frame: 36 months
Description: 412 subjects were screened and 374 subjects were enrolled in the Xenform Postmarket Surveillance Study. 228 subjects were enrolled into the Xenform arm and 146 subjects into the NTR arm. 339 subjects from the AUGS PFD Registry (64 subjects from BSC's Uphold™ LITE 522 study, 69 subjects from Acell's MatriStem® 522 study and 206 subjects from Coloplast's 522 Restorelle® study were pulled into the NTR arm for a total of 485 subjects in the NTR cohort and a total of 713 study subjects overall.
Arm/Group | Xenform | Control
All-Cause Mortality (participants affected / at risk) | 7/228 | 2/485
Serious Adverse Events (participants affected / at risk) | 20/228 | 27/485
Other Adverse Events (participants affected / at risk) | 131/228 | 312/485
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Xenform (N=228) | Control (N=485)
Cardiac Event - NEW (Cardiac disorders) | 0 (0) | 6 (6)
Cardiac Event - Worsening (Cardiac disorders) | 1 (1) | 1 (1)
Pulmonary Event, Specify - NEW (Cardiac disorders) | 1 (1) | 0 (0)
Constipation - NEW (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation - Worsening (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ileus/Bowel Obstruction (Gastrointestinal disorders) | 0 (0) | 4 (4)
Other, Specify (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Infection - Other, specify type (Infections and infestations) | 1 (1) | 4 (6)
Pelvic Infection/Abscess (Infections and infestations) | 0 (0) | 2 (2)
Pulmonary Event, Specify - NEW (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (UTI), Lower (Infections and infestations) | 0 (0) | 2 (2)
Infection - Other, specify type (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ureteral Kink/Injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Visceral Organ Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Brain Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Other, Specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Alzheimers (Nervous system disorders) | 1 (1) | 0 (0)
Mesh Exposure in Vagina (Product Issues) | 1 (1) | 0 (0)
Difficult Emptying Bladder - NEW (Renal and urinary disorders) | 3 (3) | 0 (0)
Hematoma - Retropubic (Renal and urinary disorders) | 0 (0) | 1 (1)
Stress Incontinence - Worsening (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Pelvic Pain - NEW (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Sensation of Bulge (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Other, Specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Event, Specify - Worsening (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Other, Specify (Surgical and medical procedures) | 0 (0) | 1 (1)
Bleeding (Vascular disorders) | 1 (1) | 0 (0)
Bleeding Requiring Blood Transfusion (Vascular disorders) | 2 (2) | 0 (0)
Thrombotic Event (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Xenform (N=228) | Control (N=485)
Cardiac Event - NEW (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Event - Worsening (Cardiac disorders) | 0 (0) | 1 (1)
Constipation - NEW (Gastrointestinal disorders) | 6 (6) | 12 (12)
Constipation - Worsening (Gastrointestinal disorders) | 4 (4) | 5 (5)
Fecal Incontinence - NEW (Gastrointestinal disorders) | 6 (7) | 18 (18)
Fecal Incontinence - Worsening (Gastrointestinal disorders) | 2 (2) | 6 (6)
Hematoma - Retroperitoneal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 2 (2) | 3 (3)
Ileus/Bowel Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Neuromuscular Disorder, specify type (Gastrointestinal disorders) | 0 (0) | 8 (8)
Other, Specify (Gastrointestinal disorders) | 3 (3) | 7 (7)
Cyst (General disorders) | 4 (4) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Inflammation (General disorders) | 0 (0) | 1 (1)
Neuromuscular Disorder, specify type (General disorders) | 0 (0) | 1 (1)
Other, Specify (General disorders) | 1 (1) | 2 (2)
Pain, Other (General disorders) | 1 (1) | 3 (3)
Infection - Other, specify type (Infections and infestations) | 6 (9) | 9 (10)
Other, Specify (Infections and infestations) | 0 (0) | 1 (1)
Pelvic Infection/Abscess (Infections and infestations) | 2 (2) | 3 (3)
Pulmonary Event, Specify - NEW (Infections and infestations) | 0 (0) | 2 (2)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (UTI), Lower (Infections and infestations) | 26 (39) | 118 (164)
Vaginal Infection (Infections and infestations) | 12 (14) | 16 (18)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Other, Specify (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Ureteral Kink/Injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Visceral Organ Injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Buttock Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Neuromuscular Disorder, specify type (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neoplasia, Non-Pelvic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Other, Specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuromuscular Disorder, specify type (Nervous system disorders) | 2 (2) | 6 (6)
Neurovascular Event (Nervous system disorders) | 0 (0) | 1 (1)
Other, Specify (Nervous system disorders) | 1 (1) | 0 (0)
Mesh Exposure in Vagina (Product Issues) | 2 (2) | 0 (0)
Suture Exposure in Vagina (Product Issues) | 3 (3) | 19 (20)
Other, Specify (Psychiatric disorders) | 1 (1) | 0 (0)
Difficulty Emptying Bladder - NEW (Renal and urinary disorders) | 27 (28) | 24 (25)
Difficulty Emptying Bladder - Worsening (Renal and urinary disorders) | 2 (2) | 4 (4)
Dysuria (Renal and urinary disorders) | 3 (3) | 4 (7)
Mixed Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Mixed Incontinence - Worsening (Renal and urinary disorders) | 1 (1) | 0 (0)
Mixed Urinary Incontinence (Renal and urinary disorders) | 1 (1) | 1 (1)
Other, Specify (Renal and urinary disorders) | 2 (2) | 5 (5)
Overactive Bladder (Renal and urinary disorders) | 1 (1) | 6 (6)
Stress Incontinence - NEW (Renal and urinary disorders) | 8 (8) | 6 (6)
Stress Incontinence - Worsening (Renal and urinary disorders) | 4 (4) | 21 (21)
Urge Incontinence - NEW (Renal and urinary disorders) | 14 (15) | 8 (8)
Urge Incontinence - Worsening (Renal and urinary disorders) | 8 (8) | 25 (26)
Urinary Frequency (Renal and urinary disorders) | 5 (5) | 6 (6)
Urinary Urgency (Renal and urinary disorders) | 1 (1) | 5 (5)
Weak Urinary Stream (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspareunia - NEW (De Novo) (Reproductive system and breast disorders) | 5 (6) | 11 (11)
Dyspareunia - Worsening (Reproductive system and breast disorders) | 2 (2) | 3 (3)
Hematoma - Vaginal (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Neuromuscular Disorder, specify type (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Other, Specify (Reproductive system and breast disorders) | 2 (2) | 4 (4)
Pelvic Pain - NEW (Reproductive system and breast disorders) | 17 (17) | 39 (41)
Pelvic Pain - Worsening (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Prolapse (Reproductive system and breast disorders) | 20 (21) | 88 (93)
Sensation of Bulge (Reproductive system and breast disorders) | 35 (36) | 53 (55)
Sensation of Pressure (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Vaginal Atrophy (Reproductive system and breast disorders) | 2 (2) | 3 (3)
Vaginal Bleeding, De Novo (Reproductive system and breast disorders) | 4 (4) | 9 (10)
Vaginal Discharge, Atypical (Reproductive system and breast disorders) | 2 (2) | 3 (3)
Vaginal Scarring (Reproductive system and breast disorders) | 3 (3) | 2 (2)
Vaginal Wall Dehiscence (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Vulvar Itching (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vulvar Lesion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Other, Specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lichen Sclerosus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin Condition (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Tissue Granulation (Skin and subcutaneous tissue disorders) | 9 (10) | 33 (33)
Bleeding (Vascular disorders) | 1 (1) | 1 (1)
Hematoma - Other (Vascular disorders) | 0 (0) | 1 (1)
Other, Specify (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Before publishing, Institution and Investigator shall submit copies of any proposed publication or presentation to Sponsor for review at least sixty (60) days in advance of submission for publication or presentation to a publisher or other third party. Sponsor reserves the right to delete any Confidential Information or other proprietary information of Sponsor (including trade secrets but not including Results) from the proposed publication or presentation.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/80/NCT01945580/Prot_SAP_000.pdf